CLINICAL TRIAL: NCT02884726
Title: A Phase 1 Study of the Safety and Tolerability of BMS 986148 in Subjects With Advanced and/or Metastatic Solid Tumors
Brief Title: Phase 1 Study of Mesothelin-ADC
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CA008-008
Record Dates: First submitted 2016-08-02; First posted 2016-08-31 (Estimated); Last update posted 2020-03-19 (Actual); Status verified 2020-03

CONDITIONS: Advanced Cancer

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- BMS-986148 intravenous infusion (Experimental)
  Interventions: Drug: BMS-986148

INTERVENTIONS:
Drug: BMS-986148 — Specified dose on specified days

SUMMARY:
The purpose of this study is to assess the safety and tolerability of Mesothelin-ADC in subjects with advanced and/or metastatic solid tumors.

ELIGIBILITY:
For more information regarding Bristol-Myers Squibb Clinical Trial participation, please visit www.BMSStudyConnect.com

Inclusion Criteria:

* Must have histological confirmation of advanced and/or metastatic solid

tumors which are expected to express mesothelin

* Must have received and either progressed or been intolerant to the standard treatment regimen in the advanced or metastatic setting, if such a therapy exists
* Must have measurable tumor per Response Evaluation Criteria in Solid Tumors (RECIST) or modified RECIST for malignant pleural mesothelioma
* Eastern Cooperative Oncology Group (ECOG) performance status of 0 to 1

Exclusion Criteria:

* Cancer metastases in the brain
* Uncontrolled or significant cardiovascular disease
* Moderate eye disorders
* Moderate peripheral neuropathy
* Known past or active hepatitis B or C infection

Other protocol defined inclusion/exclusion criteria could apply

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2016-10-14 (Actual); Primary Completion 2017-09-06 (Actual); Study Completion 2017-09-06 (Actual)

PRIMARY OUTCOMES:
Incidence of AEs (Adverse Events) | Day 1 to 30 days after the last dose of BMS-986148
  AEs leading to discontinuation, Death and Frequency of laboratory test toxicity grade shifting from baseline
Incidence of SAEs (Serious Adverse Events) | Day 1 to 30 days after the last dose of BMS-986148
  SAEs leading to discontinuation, Death and Frequency of laboratory test toxicity grade shifting from baseline
Grade of AEs | Day 1 to 30 days after the last dose of BMS-986148
  AE leading to discontinuation, Death and Frequency of laboratory test toxicity grade shifting from baseline
Grade of SAEs | Day 1 to 30 days after the last dose of BMS-986148
  SAEs leading to discontinuation, Death and Frequency of laboratory test toxicity grade shifting from baseline

SECONDARY OUTCOMES:
Maximum observed concentration (Cmax) | Day 1 to day 84
Time of maximum observed concentration (Tmax) | Day 1 to day 84
Area under the concentration-time curve from time zero to the time of the last quantifiable concentration [AUC(0-T)] | Day 1 to day 84
Area under the concentration-time curve in one dosing interval [AUC(TAU)] | Day 1 to day 84
Average concentration (Cavg) | Day 1 to day 84
Half life (T-half) | Day 1 to day 84
Trough observed plasma concentration (Ctrough) | Day 1 to day 84
Concentration in a dosing interval (Ctau) | Day 1 to day 84
Total body clearance (CLT) | Day 1 to day 84
Apparent volume of distribution at steady state (Vss) | Day 1 to day 84
Volume of distribution of terminal phase (Vz) | Day 1 to day 84
AUC Accumulation Index; ratio of AUC(TAU) at steady state to AUC(TAU) after the first dose (AI_AUC) | Day 1 to day 84
Cmax Accumulation Index; ratio of Cmax at steady state to Cmax after the first dose (AI_Cmax) | Day 1 to day 84
Ctau Accumulation Index; ratio of Ctau at steady state to Ctau after the first dose (AI_Ctau) | Day 1 to day 84
Response Evaluation Criteria in Solid Tumors (RECIST) | Day 1 to 30 days after the last dose of BMS-986148

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (1):
- Local Institution, Chuo-ku, Tokyo, Japan

REFERENCES:
- See also: BMS Clinical Trial Patient Recruiting — http://bms.com/studyconnect/Pages/home.aspx
- See also: Investigator Inquiry Form — http://www.bms.com/clinical_trials/Pages/Investigator_inquiry_form.aspx